CLINICAL TRIAL: NCT05624554
Title: A Phase 3, Randomized Study to Compare the Efficacy and Safety of Nemtabrutinib Versus Chemoimmunotherapy for Previously Untreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma Without TP53 Aberrations
Brief Title: A Study of Nemtabrutinib vs Chemoimmunotherapy for Participants With Previously Untreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) Without TP53 Aberrations (MK-1026-008, BELLWAVE-008)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1026-008; 2022-501481-21-00 (Registry Identifier: EU CT); MK-1026-008 (Other: MSD); U1111-1274-2574 (Registry Identifier: UTN); 2021-006593-23 (EudraCT Number)
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Cyclophosphamide; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemtabrutinib (Experimental): Administered daily via oral tablet.
  Interventions: Drug: Nemtabrutinib
- FCR or BR (Active Comparator): Investigator's choice of fludarabine plus cyclophosphamide plus rituximab (FCR) OR bendamustine plus rituximab (BR). Participants will receive either rituximab or specified approved rituximab biosimilar.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Bendamustine; Biological: Rituximab; Biological: Truxima; Biological: Ruxience; Biological: Riabni

INTERVENTIONS:
Drug: Nemtabrutinib — 65 mg administered orally daily until disease progression, unacceptable toxicity, or discontinuation criteria met.
  Other Names: MK-1026
  Arms: Nemtabrutinib
Drug: Fludarabine — 25 mg/m^2 administered via intravenous (IV) infusion on Days 1, 2, and 3 of each 28-day cycle up to 6 cycles.
  Arms: FCR or BR
Drug: Cyclophosphamide — 250 mg/m^2 administered via IV infusion on Days 1, 2, and 3 of each 28-day cycle up to 6 cycles.
  Arms: FCR or BR
Drug: Bendamustine — Administered via IV infusion on Days 1 and 2 of each 28-day cycle up to 6 cycles. The first dose is given as 70 to 90 mg/m^2. Subsequent doses may be escalated up to 90 mg/m^2, if applicable and as per local guidelines.
  Arms: FCR or BR
Biological: Rituximab — Administered as an IV infusion on Day 1 of each 28-day cycle. The initial dose is 375 mg/m^2 (cycle 1) followed by 500 mg/m^2 for remaining cycles.
  Other Names: RITUXAN®/MabThera
  Arms: FCR or BR
Biological: Truxima — Administered as an IV infusion on Day 1 of each 28-day cycle. The initial dose is 375 mg/m^2 (cycle 1) followed by 500 mg/m^2 for remaining cycles.
  Other Names: Rituximab biosimilar
  Arms: FCR or BR
Biological: Ruxience — Administered as an IV infusion on Day 1 of each 28-day cycle. The initial dose is 375 mg/m^2 (cycle 1) followed by 500 mg/m^2 for remaining cycles.
  Other Names: Rituximab biosimilar
  Arms: FCR or BR
Biological: Riabni — Administered as an IV infusion on Day 1 of each 28-day cycle. The initial dose is 375 mg/m^2 (cycle 1) followed by 500 mg/m^2 for remaining cycles.
  Other Names: Rituximab biosimilar
  Arms: FCR or BR

SUMMARY:
Researchers are looking for new ways to treat people with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL). CLL and SLL are types of blood cancer. Researchers want to know if people who take nemtabrutinib compared to those who take the standard treatments in this study will live longer without their cancer growing, spreading or returning (progression free survival).

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Confirmed diagnosis of chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL) and active disease clearly documented to have a need to initiate therapy
* Has previously untreated CLL/SLL participants without tumor protein 53 (TP53) aberrations and documented 11q status and immunoglobulin heavy chain gene (IGHV) mutational status
* The ability to swallow and retain oral medication

Exclusion Criteria:

* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Gastrointestinal dysfunction that may affect drug absorption (eg, gastric bypass surgery, gastrectomy)
* Known additional malignancy that is progressing or has required active treatment within the past 3 years, except basal cell carcinoma of skin, squamous cell carcinoma of skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potential curative therapy
* History of severe bleeding disorders
* Not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2027-05-19 (Estimated); Study Completion 2031-03-17 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Criteria 2018 as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 49 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. PD is evaluated per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria 2018 as assessed by blinded independent central review (BICR).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 94 months
  OS is defined as the time from randomization to death due to any cause.
Objective Response Rate (ORR) per iwCLL Criteria 2018 as Assessed by BICR | Up to approximately 36 months
  ORR is defined as the percentage of participants with complete response (CR), complete response with an incomplete recovery of the participant's bone marrow (CRi), nodular partial response (nPR), or Partial response (PR), per iwCLL criteria 2018 as assessed by BICR.
Duration of Response (DOR) per iwCLL Criteria 2018 as Assessed by BICR | Up to approximately 94 months
  For participants who demonstrate a CR, CRi, nPR, or PR per iwCLL criteria as assessed by BICR, DOR is defined as the time from the first documented evidence of CR, CRi, nPR, or PR that led to response until disease progression or death due to any cause, whichever occurs first.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 94 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 94 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (97):
- United States (4):
  - Highlands Oncology Group ( Site 5205), Springdale, Arkansas
  - Clermont Oncology Center ( Site 5224), Clermont, Florida
  - Hattiesburg Clinic Hematology/Oncology ( Site 5216), Hattiesburg, Mississippi
  - Medical Oncology Associates, PS ( Site 5206), Spokane, Washington
- Royal Adelaide Hospital ( Site 1105), Adelaide, South Australia, Australia
- Brazil (6):
  - Hospital Erasto Gaertner-CEPEP - Pesquisa Clínica ( Site 1317), Curitiba, Paraná
  - Hospital Amaral Carvalho-Centro de Pesquisas ( Site 1304), Jaú, São Paulo
  - A. C. Camargo Cancer Center ( Site 1318), São Paulo, São Paulo
  - Instituto Nacional de Câncer - INCA-Divisão de Pesquisa Clínica e Desenvolvimento Tecnológico HC1 ( Site 1319), Rio de Janeiro
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO-Pesquisa Clinica ( Site 1308), São Paulo
  - Hospital Paulistano-Americas Oncologia ( Site 1302), São Paulo
- Bulgaria (5):
  - Specialized Hospital for Active Treatment of Haematology Diseases ( Site 6403), Sofia, Sofia (stolitsa)
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD ( Site 6404), Plovdiv
  - Medical Centre Pratia Clinic EOOD ( Site 6406), Plovdiv
  - UMHAT "Prof. Dr. Stoyan Kirkovich"AD-Clinical Hematology ( Site 6400), Stara Zagora
  - Multriprofile Hospital for Active Treatment "Hristo Botev" ( Site 6402), Vratsa
- Chile (6):
  - IC La Serena Research ( Site 1506), La Serena, Coquimbo Region
  - Centro de Estudios Clínicos SAGA-CECSAGA ( Site 1509), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 1500), Santiago, Region M. de Santiago
  - Clínica Inmunocel ( Site 1511), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 1503), Temuco, Región de la Araucanía
  - Biocenter ( Site 1507), Concepción, Región del Biobío
- China (23):
  - Peking University Third Hospital ( Site 1602), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 1605), Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital ( Site 1609), Chongqing, Chongqing Municipality
  - Southern Medical University Nanfang Hospital-Department of Hematopathology ( Site 1607), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center ( Site 1608), Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University ( Site 1625), Guiyang, Guizhou
  - Hainan General Hospital ( Site 1603), Haikou, Hainan
  - Henan Cancer Hospital-hematology department ( Site 1613), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 1619), Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 1618), Wuhan, Hubei
  - Xiangya Hospital Central South University-Hematology department ( Site 1616), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 1615), Changsha, Hunan
  - The First Affiliated Hospital of Soochow University-hematology department ( Site 1612), Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 1614), Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital ( Site 1628), Nanchang, Jiangxi
  - The First Hospital of Jilin University-Hematology ( Site 1621), Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 1617), Xi'an, Shaanxi
  - Shaanxi provincial people's hospital ( Site 1626), Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center ( Site 1606), Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital ( Site 1629), Taiyuan, Shanxi
  - Institute of hematology&blood disease hospital ( Site 1600), Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital-lymphoma ( Site 1604), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University-Hematology ( Site 1611), Hangzhou, Zhejiang
- Colombia (4):
  - Clini Salud ( Site 1700), Envigado, Antioquia
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 1707), Medellín, Antioquia
  - Sociedad De Oncologia Y Hematologia Del Cesar-Oncology ( Site 1704), Valledupar, Cesar Department
  - Oncologos del Occidente ( Site 1706), Pereira, Risaralda Department
- Denmark (4):
  - Aarhus Universitetshospital, Skejby-Blodsygdomme ( Site 1902), Aarhus, Central Jutland
  - Aalborg Universitetshospital, Syd ( Site 1901), Aalborg, North Denmark
  - Odense Universitetshospital ( Site 1900), Odense C, Region Syddanmark
  - Vejle Sygehus ( Site 1903), Vejle, Region Syddanmark
- Guatemala (3):
  - MEDI-K ( Site 2401), Guatemala City
  - CELAN,S.A ( Site 2403), Guatemala City
  - Oncomedica ( Site 2402), Guatemala City
- Queen Mary Hospital ( Site 2500), Hksar, Hong Kong
- Hungary (3):
  - Fejér Megyei Szent György Egyetemi Oktató Kórház ( Site 2609), Székesfehérvár, Fejér
  - Heves Vármegyei Markhot Ferenc Oktatókórház és Rendelőintézet ( Site 2608), Eger, Heves County
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókór-Haematológia osztály ( Site 2602), Nyíregyháza, Szabolcs-Szatmár-Bereg
- Hospital of Lithuanian University of Health Sciences Kauno klinikos-Oncology and Hematology ( Site 3100), Kaunas, Kaunas County, Lithuania
- Malaysia (2):
  - Hospital Sultanah Aminah ( Site 3203), Johor Bahru, Johor
  - Hospital Ampang ( Site 3202), Ampang, Selangor
- Mexico (4):
  - Centro de Infusion Superare ( Site 3314), Mexico City, Mexico City
  - Health Pharma Professional Research S.A. de C.V: ( Site 3301), Mexico City, Mexico City
  - Centro de Investigacion Clinica Chapultepec ( Site 3309), Morelia, Michoacán
  - Oaxaca Site Management Organization ( Site 3313), Oaxaca City
- Poland (6):
  - Uniwersytecki Szpital Kliniczny nr 1 w Lublinie ( Site 3710), Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Układu Chłonnego ( Site 3701), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Hematologii i Transplantologii ( Site 3702), Gdansk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice ( Site 3705), Katowice, Silesian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej MSWiA z Warmi-Oddzial Kliniczny Hematologii ( Site 3704), Olsztyn, Warmian-Masurian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Hematologii i Transplantacji S ( Site 3711), Kielce, Świętokrzyskie Voivodeship
- Romania (3):
  - Spitalul Clinic Colțea ( Site 4000), Bucharest, București
  - Spitalul Clinic Colțea ( Site 4001), Bucharest, București
  - Institutul Oncologic Cluj ( Site 4002), Cluj-Napoca
- Singapore (2):
  - National Cancer Centre Singapore ( Site 4200), Singapore, Central Singapore
  - Tan Tock Seng Hospital ( Site 4202), Singapore, Central Singapore
- South Africa (5):
  - Netcare Pretoria East Hospital-Albert Alberts Stem Cell Transplant Centre ( Site 4401), Centurion, Gauteng
  - Wits Clinical Research ( Site 4403), Johannesburg, Gauteng
  - Groote Schuur Hospital-Clinical Haematology ( Site 4400), Cape Town, Western Cape
  - Haemalife ( Site 4407), Kuilsriver, Western Cape
  - Constantiaberg Haematology ( Site 4408), Plumstead, Western Cape
- Taiwan (3):
  - Chang Gung Memorial Hospital at Kaohsiung-Division of Hematology and Oncology ( Site 4700), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 4701), Tainan
  - National Taiwan University Hospital ( Site 4704), Taipei
- Turkey (Türkiye) (5):
  - Mega Medipol-Hematology ( Site 4904), Stanbul, Istanbul
  - Namik Kemal University Medical Faculty-Hematology ( Site 4912), Suleymanpasa, Tekirdas
  - Ankara Universitesi Tip Fakultesi Hastanesi-hematology ( Site 4913), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi ( Site 4906), Istanbul
  - Ege Universitesi Hastanesi ( Site 4902), Izmir
- Ukraine (6):
  - MNPE ClinCenter of Oncology,Hematology,Transplantology and Palliative Care of CherkasyRegCouncil ( Site 5106), Cherkassy, Cherkasy Oblast
  - Communal non-profit enterprise "Regional clinical hospital o-Hematology Department ( Site 5113), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Nonprofit Organization National Cancer Institute ( Site 5103), Kyiv, Kyivska Oblast
  - Institute of Blood Pathology and Transfusion Medicine of National Aсademy of Medical Sciences of Ukr ( Site 5105), Lviv, Lviv Oblast
  - SI National Research Center of Radiation Medicine, Hematology, Oncology ( Site 5101), Kyiv
  - Public Non-Profit Enterprise Kyiv City Clinical Hospital #9 -Hematology department #1 ( Site 5111), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26189&tenant=MT_MSD_9011